CLINICAL TRIAL: NCT01722058
Title: A Phase I In-Vivo Colon Protocol for Detection of Neoplasia in the Digestive Tract (U54)
Brief Title: A Phase I In-Vivo Peptide Applied in the Right Colon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Missy Tuck, Project Manager, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00068009
Record Dates: First submitted 2012-10-30; First posted 2012-11-06 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Colon Lesions
Keywords: peptide; colon; flat lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peptide application (Experimental)
  Interventions: Drug: Peptide application

INTERVENTIONS:
Drug: Peptide application
  Other Names: Colon KCC Heptapeptide (5-FITC-labeled peptide)

SUMMARY:
You are invited to participate in a research study to develop new ways to look for abnormal areas/tissues of the colon. The current endoscopes used to look at the colon are very good, but if the area doesn't look different to the naked eye, then the endoscope can't improve on that. We are looking at using special fluorescent stains in addition to special endoscopes designed to see abnormal areas that are not obvious to the naked eye. Currently specialized microscopes and fluorescent stains are used in clinical laboratories but it takes several days of processing to get results. It may be very helpful to look for areas to sample for abnormal tissue during the endoscopy procedure.

You are being asked to let us spray a "fluorescent peptides" into your right colon. Peptides are small chains of amino acids (the building blocks that make up proteins) linked together. Our peptide is a chain of 7 amino acids attached to a fluorescent dye called FITC (like the one used by your eye doctor).

We have prepared this special "fluorescent peptide" to target and bind to any abnormal areas if present, and "glow" when a special light is used. In this study, we will apply the special fluorescent peptide by a spray catheter to your right colon to asses for safety. The colonoscope used in this study is the usual colonoscope used and is not able to see the fluorescence.

This is a phase 1 study. This means that this is the first time we have used this kind of "fluorescent peptide" in people. The Food and Drug Administration (FDA) has not approved this agent, but is allowing us to test it in this study. The goal of this study is to see if there are any side effects from using the peptide. We have used a similar peptide that we've developed for the esophagus in over 40 patients without any side effects.

This is the first test of this agent, so it won't be used to change how colonoscopy is done.

DETAILED DESCRIPTION:
The goal of this research is to develop the use of fluorescence-labeled peptides (Colon KCC) that affinity bind to pre-cancerous mucosa in the digestive tract for use as an imaging agent to aid in the early detection of colon cancer. Currently colon cancer prevention is achieved by endoscopic evaluation and removal of pre-malignant lesions (adenomatous polyps) by endoscopic resection and biopsy. Standard endoscopy uses white light illumination and is only able to detect pre-cancerous tissue that has abnormal architectural features, such as a polyp or mass. However, pre-cancerous lesions can also be flat in appearance and visually indistinct from normal tissue; such as in the case of chronic ulcerative colitis and / or some right-sided polyps.

Furthermore, flat and depressed lesions, which are more difficult to detect in white light colonoscopy, may represent over 25% of all pre-malignant lesions and may confer a higher risk for malignancy. Integration of molecular probes that home in to diseased tissues with high resolution imaging instruments could greatly improve the diagnostic accuracy for missed lesions of both polypoid and non-polypoid morphology, including the often fatal 'right-sided ' adenomas.

Endoscopic imaging with the use of fluorescent-labeled probes is a promising method for achieving greater specificity, spatial localization and higher image contrast in the detection of neoplastic lesions. This study is a 'first-in-humans' test of the safety of the topically applied peptide.

A Phase I study of the safety of a topically-administered fluorescent heptapeptide for detecting neoplastic areas of the colon is proposed. The study will test the safety of administering this agent to human subjects undergoing clinically-indicated colonoscopy. Safety is defined as the occurrence of adverse events after the administration of topical fluorescence-labeled peptides to the surface of intra-colonic mucosa.

ELIGIBILITY:
The inclusion criteria for this proposed clinical study are:

* Subjects who are scheduled for outpatient colonoscopy.
* All subjects who are medically cleared for the procedure (e.g. washout for anticoagulants, comorbidities) who meet the inclusion/exclusion will be included. Standard practice guidelines for safely proceeding with the procedure will be sufficient for our study
* Adults aged 18 years to 100
* Willing and able to sign informed consent
* Willing and able to get the repeat clinical labs
* The effects of the Colon KCC Heptapeptide (labeled with 5-FITC) on the developing human fetus are unknown. For this reason, women of child-bearing potential must have a negative pregnancy test on the day of the procedure to receiving the Colon KCC Heptapeptide (5-FITC-labeled peptide) agent or be post-menopausal. Post-menopausal women are defined as post-hysterectomy, or over 40 and at least 18 months without menses and not on birth-control.

The exclusion criteria for this proposed clinical study are:

* Subjects with known allergy or negative reaction to fluorescein or derivatives.
* Subjects on active chemotherapy or radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Application of peptide to 25 subjects undergoing colonoscopy | 6 months
  To evaluate the safety of topically administered fluorescence-labeled peptides to the surface of intra-colonic mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kim Turgeon, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States